CLINICAL TRIAL: NCT00444977
Title: Enhancing Oral Health Care Use by HIV-Positives
Brief Title: Enhancing Oral Health Care Use by HIV Positive Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lisa Metsch (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor-Investigator, Lisa Metsch, Stephen Smith Professor of Sociomedical Sciences and Chair, Department of Sociomedical Sciences, Columbia University
Organization: Columbia University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AAAK3159; R01DE015523 (NIH)
Record Dates: First submitted 2007-03-06; First posted 2007-03-08 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Oral Health Care; HIV Infections; Mouth Diseases
Keywords: HIV positive persons; Not received oral health care in the preceding 12 months.; treatment naive; treatment experienced
MeSH Terms: conditions — HIV Infections; Mouth Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case-management linkage intervention (Experimental): The intervention represents a brief, "real world" intervention that could easily be adopted by HIV care clinics to facilitate linkage and increase use of oral services by their HIV+ patients (if shown to be effective). We are seeking to compare this intervention to usual practice in these clinics.
  Interventions: Behavioral: Case-management linkage intervention
- Standard of Care (No Intervention): Subjects will receive standard of care services.

INTERVENTIONS:
Behavioral: Case-management linkage intervention — dental care
  Arms: Case-management linkage intervention

SUMMARY:
The purpose of this study is to investigate the efficacy of a case management linkage intervention designed to increase utilization of oral health care services among HIV+ individuals enrolled in HIV primary care that have not seen a dental provider in the preceding twelve months.

DETAILED DESCRIPTION:
Recent national studies demonstrate that oral health is one of the highest unmet health needs for HIV-positive (HIV+) individuals, although it is recognized as playing a less critical role in the medical management of HIV/AIDS. Social and economic factors have contributed to less than optimal use of oral health services for HIV+s in the United States. According to recent data, from Miami-Dade County, Florida, only 24% of HIV+s served by Ryan White-funded medical clinics had obtained oral health services in the past 12 months.

To address the underutilization of oral health care services, we propose to develop, implement, and evaluate an intervention to assist low-income HIV+s in obtaining access to oral health services as well as increase appropriate utilization of these services. The case management intervention is adapted from an intervention that had been previously tested in a CDC-funded, multi-site study designed to link recently diagnosed HIV+s to primary medical care.

A two-arm randomized trial among HIV+ individuals who are currently enrolled in HIV primary medical care, but not receiving oral health care, will be conducted to test the intervention. The two arms will consist of a case management intervention and standard-of-care. Participants will be assessed at baseline and at 6, 12 and 18 months after baseline to document their utilization of oral health services. An interdisciplinary team of behavioral and clinical research scientists with experience in developing and evaluating health care and prevention intervention targeting low income, HIV+s will conduct this research.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years and older
* Documented HIV infection
* Currently in medical care (defined as having seen an HIV primary care provider in the previous six months)
* Eligible for Ryan White title I funding
* Plans to remain in Miami for the next 24 months
* Provide the name of two verifiable locator persons

Exclusion Criteria:

* Persons not meeting the inclusion criteria as delineated above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2005-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
dental visit and screening resulting from case management | 6, 12 and 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa R Metsch, PhD, Principal Investigator — Columbia University
Locations (1):
- University of Miami, Miami, Florida, United States